CLINICAL TRIAL: NCT03071107
Title: Frailty Intervention Trial in End-Stage Patients on Dialysis: A Feasibility Study
Brief Title: Frailty Intervention Trial in End-Stage Patients on Dialysis
Acronym: FITNESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adnan Sharif (Other)
Responsible Party: Sponsor-Investigator, Adnan Sharif, Chief Investigator, University Hospital Birmingham NHS Foundation Trust
Organization: University Hospital Birmingham NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FITNESS
Record Dates: First submitted 2017-02-25; First posted 2017-03-06 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Hemodialysis Complication; Nutritional Deficiency; Physical Activity
MeSH Terms: conditions — Malnutrition; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-disciplinary intervention arm (Active Comparator): Multi-disciplinary intervention on frailty parameters including input from dietitian, physiotherapist and medical team
  Interventions: Behavioral: Multi-disciplinary intervention
- Control arm (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Multi-disciplinary intervention — Participants in the intervention group will receive a multifactorial, interdisciplinary, treatment program intended to target pre-frailty for a 4-month period following randomization (physical meetings at 2-monthly time points with telephone consultations between meetings). The interventions will be individually tailored to each participant based on their frailty characteristics at baseline and amended if other problems are identified during the intervention program. This intervention team will consist of a renal dietitian and physiotherapist, both of whom will be trained and accredited in behavioural therapy intervention skills, and will focus on improving nutritional status and physical strength through resistance exercise training. They will be supported by a Clinical Research Fellow who will provide additional medical assessment to determine any reversible medical causes of frailty.
  Arms: Multi-disciplinary intervention arm

SUMMARY:
The proposed investigation for this study aims to; 1) understand the prevalence and outcomes associated with frailty among haemodialysis patients; 2) ascertain the best frailty assessment tool for haemodialysis patients, and; 3) design a clinical study to explore the feasibility of facilitating, recruiting and executing a multi-disciplinary clinical and psychological intervention to improve frailty status among haemodialysis patients.

Work package 1: Firstly, there is a need to understand the prevalence and spectrum of frailty in a UK haemodialysis cohort and what impact frailty has for haemodialysis patients. To investigate this, the investigators will approach every patient on haemodialysis within the local catchment of haemodialysis units and, after informed consent, clinically phenotype their frailty status (pre- and post-haemodialysis for calculation of variability). The frailty phenotyping will encompass a number of frailty assessments (including the Edmonton Frail Scale, Clinical Frailty Scale from Rookwood score and Fried Frailty scale) to identify the ideal frailty assessment tool. All patients in this observational cohort study will be prospectively monitored for clinical/biochemical outcomes using an informatics-based approach for up to 60 months.

Work package 2: Building upon the work conducted in work package 1, work package 2 will aim to recruit 50 patients clinically phenotyped with pre-frailty from work package 1 into a feasibility study exploring a multi-disciplinary intervention to improve frailty status. Eligible patients, after informed consent, will be randomised into active or passive intervention. The active intervention will involve a dietitian and physiotherapist who have been trained and accredited with cognitive behavior intervention, utilising established behavioral intervention frameworks, to deliver a multi-disciplinary clinical intervention targeting multiple components of frailty.

The FITNESS project will therefore answer some important unanswered questions regarding frailty among the haemodialysis population and help in the design of a large multi-disciplinary intervention study if deemed feasible.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis

Exclusion Criteria:

* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of frailty intervention study in haemodialysis patients | 6-months
  Feasibility of undertaking a full scale clinical intervention trial targeting frail haemodialysis patients

SECONDARY OUTCOMES:
Change in frailty status | 6-months
  Change in frailty score between baseline and end of study
Mortality | 6-months
  Difference in mortality episodes between randomised arms
Hospitalisation | 6-months
  Difference in episodes of hospitalisation between randomised arms

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson BM, Qasim M, Correa G, Evison F, Gallier S, Ferro CJ, Jackson TA, Sharif A. A clinical frailty scale obtained from MDT discussion performs poorly in assessing frailty in haemodialysis recipients. BMC Nephrol. 2023 Mar 30;24(1):80. doi: 10.1186/s12882-023-03126-0. PMID 36997856
- [Derived] Anderson BM, Wilson DV, Qasim M, Correa G, Evison F, Gallier S, Ferro CJ, Jackson TA, Sharif A. Ultrasound quadriceps muscle thickness is variably associated with frailty in haemodialysis recipients. BMC Nephrol. 2023 Jan 18;24(1):16. doi: 10.1186/s12882-022-03043-8. PMID 36653750
- [Derived] Anderson BM, Dutton M, Day E, Jackson TA, Ferro CJ, Sharif A. Frailty Intervention Trial iN End-Stage patientS on haemodialysis (FITNESS): study protocol for a randomised controlled trial. Trials. 2018 Aug 24;19(1):457. doi: 10.1186/s13063-018-2842-x. PMID 30143028